CLINICAL TRIAL: NCT00821119
Title: A Randomized Controlled Trial of Nasal Intermittent Positive Pressure Ventilation Versus Nasal Continuous Positive Pressure as a Primary Mode for Respiratory Distress Syndrome in Preterm Infants
Brief Title: Trial of Non Invasive Ventilation for Respiratoy Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Jucille do Amaral Meneses, Jucille Meneses Md PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMIP123
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Prematurity; Respiratory Distress Syndrome
Keywords: non invasive ventilation; mechanical ventilation; pulmonary morbidity; preterm infant; Respiratory distress syndrome; nasal intermittent positive pressure; nasal continuous positive pressure; bronchopulmonary dysplasia
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NCPAP (Active Comparator): preterm infants with nasal positive pressure ventilation as a primary mode of respiratory support in preterm infants with respiratory distress syndrome will be compared to preterm infants with nasal intermittent positive pressure ventilation
  Interventions: Device: nasal intermittent positive pressure ventilation
- NIPPV (Experimental): preterm with nasal intermittent positive pressure ventilation as a primary mode of respiratory support in preterm infants with respiratory distress syndrome
  Interventions: Device: nasal intermittent positive pressure ventilation

INTERVENTIONS:
Device: nasal intermittent positive pressure ventilation — Nasal intermittent positive airway pressure will be compared are the nasal continuous positive pressure as an initial ventilatory mode in preterm infants with respiratory distress syndrome
  Other Names: NIPPV

SUMMARY:
The purpose of this study is to evaluate the hypothesis that nasal intermittent positive pressure(NIPP), used as a primary mode of ventilation in preterm infants with RDS, will decrease the need for conventional endotracheal ventilation when compared to nasal continuous positive airway pressure.(NCPAP)

DETAILED DESCRIPTION:
Respiratory distress syndrome(RDS) and its sequelae, bronchopulmonary dysplasia(BPD) are complications of prematurity.The pathogenesis of BPD is multifactorial and one of the most important risk factors is the ventilator-induced lung injury caused by invasive respiratory support.

The two modes of non-invasive ventilation, NIPP and specially NCPAP, have been used frequently in the respiratory care of preterm infants in neonatal units.NCPAP is currently a common practice for the treatment of RDS . NIPP has been found to be more effective than NCPAP in apnea of prematurity and immediately after extubation in preterm infants,decreasing the need of endotracheal ventilation.

Alternative techniques of non-invasive ventilation has been suggested in some studies to decrease respiratory morbidities associated with prematurity.This non-invasive approach could be used initially as a primary mode of ventilation for infants with RDS in a effort to decrease lung injury and BPD.Studies are needed to compare the effectiveness of these therapies.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with RDS
* assigned to non invasive ventilation

Exclusion Criteria:

* preterm on endotracheal ventilation
* severe congenital pulmonary or cardiovascular malformation

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao Guilherme B Alves, PhD, Study Director — Instituto Materno Infantil Prof. Fernando Figueira
Locations (2):
- Brazil (2):
  - Maternal Infant Institute Prof Fernando Figueira, Recife, Pernambuco
  - Instituto materno Infantil Fernando Figueira, Recife, Pernambuco

REFERENCES:
- [Background] Ambalavanan N, Carlo WA. Ventilatory strategies in the prevention and management of bronchopulmonary dysplasia. Semin Perinatol. 2006 Aug;30(4):192-9. doi: 10.1053/j.semperi.2006.05.006. PMID 16860159
- [Background] Bancalari E, del Moral T. Continuous positive airway pressure: early, late, or stay with synchronized intermittent mandatory ventilation? J Perinatol. 2006 May;26 Suppl 1:S33-7; discussion S43-5. doi: 10.1038/sj.jp.7211471. PMID 16625223
- [Background] Van Marter LJ, Allred EN, Pagano M, Sanocka U, Parad R, Moore M, Susser M, Paneth N, Leviton A. Do clinical markers of barotrauma and oxygen toxicity explain interhospital variation in rates of chronic lung disease? The Neonatology Committee for the Developmental Network. Pediatrics. 2000 Jun;105(6):1194-201. doi: 10.1542/peds.105.6.1194. PMID 10835057
- [Background] Bhandari V, Gavino RG, Nedrelow JH, Pallela P, Salvador A, Ehrenkranz RA, Brodsky NL. A randomized controlled trial of synchronized nasal intermittent positive pressure ventilation in RDS. J Perinatol. 2007 Nov;27(11):697-703. doi: 10.1038/sj.jp.7211805. Epub 2007 Aug 16. PMID 17703184
- [Background] De Paoli AG, Davis PG, Lemyre B. Nasal continuous positive airway pressure versus nasal intermittent positive pressure ventilation for preterm neonates: a systematic review and meta-analysis. Acta Paediatr. 2003;92(1):70-5. doi: 10.1111/j.1651-2227.2003.tb00472.x. PMID 12650303
- [Background] Santin R, Brodsky N, Bhandari V. A prospective observational pilot study of synchronized nasal intermittent positive pressure ventilation (SNIPPV) as a primary mode of ventilation in infants > or = 28 weeks with respiratory distress syndrome (RDS). J Perinatol. 2004 Aug;24(8):487-93. doi: 10.1038/sj.jp.7211131. PMID 15141265
- [Background] Manzar S, Nair AK, Pai MG, Paul J, Manikoth P, Georage M, Al-Khusaiby SM. Use of nasal intermittent positive pressure ventilation to avoid intubation in neonates. Saudi Med J. 2004 Oct;25(10):1464-7. PMID 15494823
- [Background] Kugelman A, Feferkorn I, Riskin A, Chistyakov I, Kaufman B, Bader D. Nasal intermittent mandatory ventilation versus nasal continuous positive airway pressure for respiratory distress syndrome: a randomized, controlled, prospective study. J Pediatr. 2007 May;150(5):521-6, 526.e1. doi: 10.1016/j.jpeds.2007.01.032. PMID 17452229
- [Derived] Meneses J, Bhandari V, Alves JG, Herrmann D. Noninvasive ventilation for respiratory distress syndrome: a randomized controlled trial. Pediatrics. 2011 Feb;127(2):300-7. doi: 10.1542/peds.2010-0922. Epub 2011 Jan 24. PMID 21262883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The started study date of recruitment was March 2008 in a single center. One of the biggest hospital in the northeast of brazil with an inborn tertiary NICU
Pre-assignment Details: Infants were excluded for any of the following reasons: major congenital anomalies, presence of cardiovascular instability, intubation at admission to the NICU, consent not provided or refused and unavailability of a ventilator. there were 423 eligible infants and 223 excluded, 200 participated in the study
Groups:
- Nasal Continuous Positive Airway Pressure (NCPAP): Continuous nasal positive airway pressure as a mode of respiratory support in preterm infants with respiratory distress syndrome from birth up to 72 hours of life. Infants randomized to the NCPAP group were initiated on a pressure of 5 - 6 cm H2O and a flow of 8 - 10L/m by an underwater seal (Bubble CPAP system, Intermed Inc., Sao Paulo, Brazil). Short binasal prongs were used and settings were adjusted to target a SpO2 between 88 - 92%.
- Nasal Intermittent Positive Pressure Ventilation (NIPPV): Nasal intermittent positive pressure ventilation as a mode of respiratory support in preterm infants with respiratory distress syndrome from birth up to 72 hours of life.We used a time-cycle, pressure-limited and continuous flow neonatal ventilator (Inter Neo, Intermed Inc., Sao Paulo, Brazil) for infants assigned to the NIPPV group, in the non-synchronized mode. The initial settings were: frequency of 20 to 30 breaths per minute, peak inspiratory pressure (PIP) of 15 to 20 cm H2O, peak end expiratory pressure (PEEP) of 4 - 6 cm H2O, inspiratory time (Ti) of 0.4 - 0.5 s and a flow of 8 - 10L/m.Short binasal prongs were used and settings were adjusted to target a SpO2 between 88 - 92%.
Period: Overall Study
Arm/Group | Nasal Continuous Positive Airway Pressure (NCPAP) | Nasal Intermittent Positive Pressure Ventilation (NIPPV)
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 - NCPAP: preterm infants with nasal continuous positive pressure as the mode of respiratory support
- 2- NIPP: preterm with nasal intermittent positive pressure ventilation as a primary mode of respiratory support
- Total: Total of all reporting groups
Arm/Group | 1 - NCPAP | 2- NIPP | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 100 | 200
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: weeks of gestation] | 30.1 (2.3) | 29 (1.6) | 30 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 49 | 100
  Male | 49 | 51 | 100
Region of Enrollment [Number; unit: participants]
  Brazil | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Need for Endotracheal Ventilation in the First 72 hs of Life
Description: number of participants that needed endotracheal ventilation (failed non invasive ventilation) in the first 72 hours of life
Time Frame: first 72 hs of life
Population: 40 - 45% of our previous preterm infants on NCPAP for RDS needed intubation and mechanical ventilation within the first 72h of life. We estimated a 20% absolute reduction in the need of using ETT ventilation with the early use of NIPPV. A sample size of 100 infants per group was calculated with a power of 80% and an alpha error of 5%.
Measure: Number; unit: participants
Groups:
- NCPAP: preterm infants with nasal continuous positive pressure as the mode of respiratory support
- NIPPV: preterm infants with nasal intermittent positive pressure ventilation as a primary mode of respiratory support
Arm/Group | NCPAP | NIPPV
Number analyzed (Participants) | 100 | 100
participants | 34 (0) | 25 (0)
Statistical Analysis 1: Comparison: NCPAP vs NIPPV; Based on previous data from our NICU, 40 - 45% of our preterm infants administered early NCPAP for RDS needed intubation and mechanical ventilation within the first 72h of life. We estimated a 20% absolute reduction in the need of using ETT ventilation with the early use of NIPPV. A sample size of 100 infants per group was calculated with a power of 80% and an alpha error of 5%. The analysis was performed according to the intention-to-treat principle; Test type: Superiority or Other; p < 0.05, risk ratio (RR); Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.48 to 1.14], Standard Error of Mean 0.16

2. Primary Outcome: Mechanical Ventilation Within the First 72h of Life in the Two Study Groups.(NIPPV vs NCPAP)
Description: The primary outcome of the study was the need for intubation within the first 72 hours (h) of life.The need for intubation was made by the attending neonatologist, according to the strict protocol of intubation for ventilation, used in the neonatal Unit
Time Frame: first 3 days of life(72hours)
Population: We estimated a 20% absolute reduction in the need of using endotraqueal ventilation with the early use of NIPPV. A sample size of 100 infants per group was calculated with a power of 80% and an alpha error of 5%.
Measure: Number; unit: participants
Groups:
- NCPAP: Preterm infants with nasal continuous positive pressure as the mode of respiratory support.Infants randomized to the NCPAP group were initiated on a pressure of 5 - 6 cm H2O and a flow of 8 - 10L/m by an underwater seal (Bubble CPAP system, Intermed Inc., Sao Paulo, Brazil). Short binasal prongs were used and settings were adjusted to target a SpO2 between 88 - 92%.
- NIPPV: Preterm infants with nasal intermittent positive pressure ventilation as a primary mode of respiratory support. These infants were treated with time-cycle, pressure-limited and continuous flow neonatal ventilator (Inter Neo, Intermed Inc., Sao Paulo, Brazil) for infants assigned to the NIPPV group, in the non-synchronized mode. The initial settings were: frequency of 20 to 30 breaths per minute, peak inspiratory pressure (PIP) of 15 to 20 cm H2O, peak end expiratory pressure (PEEP) of 4 - 6 cm H2O, inspiratory time (Ti) of 0.4 - 0.5 s and a flow of 8 - 10L/m.Short binasal prongs were used and settings were adjusted to target a SpO2 between 88 - 92%.
Arm/Group | NCPAP | NIPPV
Number analyzed (Participants) | 100 | 100
participants | 34 [0.48 to 1.14] | 25 [0.48 to 1.14]
Statistical Analysis 1: Comparison: NCPAP vs NIPPV; Based on previous data from our NICU, 40 - 45% of our preterm infants administered early NCPAP for RDS needed intubation and mechanical ventilation within the first 72h of life. We estimated a 20% absolute reduction in the need of using ETT ventilation with the early use of NIPPV. A sample size of 100 infants per group was calculated with a power of 80% and an alpha error of 5%; Test type: Superiority or Other; p = 0.05, risk ratio (RR); Risk Ratio (RR) = 0.70, 95% CI 2-sided [0.48 to 1.14], Standard Error of Mean 0.16

3. Secondary Outcome: Bronchopulmonary Dysplasia
Description: The incidence of bronchopulmonary dysplasia was calculated based on the number of infants surviving to 36 weeks postmenstrual age and diagnosed with bronchopulmonary dysplasia, according to the definiton of bronchopulmonary dysplasia currently used in the neonatal Unit.
Time Frame: at 36 weeks gestational age
Population: The number of preterm infants surviving to 36 weeks postmenstrual age were eligible for analysis
Measure: Number; unit: participants
Arm/Group | NCPAP | NIPPV
Number analyzed (Participants) | 80 | 83
participants | 20 | 22
Statistical Analysis 1: Comparison: NCPAP vs NIPPV; The study was not powered for this outcome. However this analysis was done with this limitation; Test type: Superiority or Other; p < 0.05, risk ratio (RR); Risk Ratio (RR) = 1.06, 95% CI 2-sided [0.62 to 1.78], Standard Error of Mean 0.18

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during 2 years
Arm/Group | 1 - NCPAP | 2- NIPP
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No